CLINICAL TRIAL: NCT06109610
Title: A Randomized Control Trial of Cognitive Behavioral Therapy on Adherence and Depression (CBT-AD) Among HIV/AIDS Patients on Follow up at Mattu Karl and Bedele Hospital, 2019
Brief Title: Cognitive Behavioral Therapy on Adherence and Depression (CBT-AD) Among HIV/AIDS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mattu University (Other)
Responsible Party: Principal Investigator, Zakir Abdu, Assistant Professor of Psychiatry, Mattu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHS/19/2019
Record Dates: First submitted 2023-10-17; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Depression; Medication Adherence
MeSH Terms: conditions — Depression; Medication Adherence | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Taking Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Control group (No Intervention): Do not taking Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The treatment will be offered to participants free of charge. Cognitive Behavioral Therapy (CBT) sessions will be delivered in a group therapy format and the sessions will be offered in successive weeks. The protocol will be then administered to the intervention group (in 8 groups over a period of six months, eight sessions, each of 30 minutes' length).
  Arms: Intervention group

SUMMARY:
Depression is highly comorbid with HIV/ AIDS and is associated with worse poor adherence to antiretroviral therapy (ART), and potentially to long-term immune functioning. Cognitive behavioral therapy may solve these problem.

DETAILED DESCRIPTION:
Depression is highly comorbid with HIV/ AIDS and is associated with worse poor adherence to antiretroviral therapy (ART), and potentially to long-term immune functioning. Poor adherence decreases the benefits of ART as well as chances of prolonged survival. An intervention that integrates CBT for depression with a cognitive behavioral approach to adherence counseling (cognitive behavioral therapy intervention for adherence and depression (CBT-AD)) has been found to be effective in improving adherence and reducing depression in PLWH.

ELIGIBILITY:
Inclusion Criteria:

* PLWHA who were 18 years old and above were included in the study

Exclusion Criteria:

* PLWHA who were previously took CBT and participants with acute physical or mental disturbances were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
The mean score of Depression will change after intervention | Through study completion, an average of 1 yea
  Depression is measured by Patient Health Questionnaire (PHQ-9) Depression Scale. The minimum value is 0 and the maximum value is 27. The higher score mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Zakir Abdu, MSc, Principal Investigator — Mattu Universitry; Mohammedamin Hajure, MSc, Study Chair — Mattu University
Locations (1):
- Mattu University, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Any qualified researchers could get the data from principal investigator at any time